CLINICAL TRIAL: NCT05104710
Title: Intermuscular Coherence: A Biomarker for Early Diagnosis and Follow-up of ALS
Brief Title: Intermuscular Coherence as a Biomarker for ALS
Acronym: ALS-IMC
Status: Recruiting | Type: Observational
Sponsor: University of Chicago (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Massachusetts General Hospital (Other); Washington University School of Medicine (Other); University of California, Irvine (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB20-1478; 1R01NS116262-01A1 (NIH)
Record Dates: First submitted 2021-10-21; First posted 2021-11-03 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (3):
- AIM 1: Hypothesis: IMC-βγ can help to differentiate between ALS and mimic diseases at initial presentation.
  Patients who present to a neuromuscular clinic with symptoms that might be from ALS but for whom a diagnosis is not yet known, will be studied. Measurements of intermuscular coherence will be made using surface electrodes. A standard neurological examination and questionnaire about ALS symptoms will be completed. No interventions will be made. A patient's final diagnosis will be determined using standard-of-care testing. Six months after initial IMC measurement, a determination will be made whether the IMC predicted the diagnosis of ALS.
- AIM 2: Hypothesis: Characterization of demographic-specific distributions will improve the specificity of IMC-βγ for ALS.
  To optimize cutoff values for abnormal IMC, IMC-βγ will be measured in neurotypical controls across a range of age, race, ethnicity, and sexes.
- AIM 3: Hypothesis: IMC-βγ will decrease with disease progression.
  Because IMC-βγ measures functional input from motor neurons in the brain, it should decrease as these neurons are lost. IMC will be measured sequentially about every 3 months in patients with ALS, and will be compared to measures of clinical progression.

SUMMARY:
The specific aims of this study are to:

1. Determine if a painless and quick measurement of muscle activity using surface electrodes can help with the diagnosis of ALS. Specifically, we ask if a measure of intermuscular coherence (IMC-βγ), when added to current diagnostic criteria (Awaji criteria), can differentiate ALS from mimic diseases more accurately and earlier than currently possible.
2. Characterize IMC-βγ in neurotypical subjects by age, sex, race, and ethnicity.
3. Follow a cohort of ALS patients longitudinally to determine if IMC-βγ changes with ALS disease progression and whether such changes correlate with functional and clinical scores, or survival.

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis (ALS) is a fatal neurodegenerative disease caused by neuronal death in the motor system, both in the brain and spinal cord. It results in progressive weakness throughout the body, and typically leads to respiratory failure 3-5 years after symptom onset. Therapy initiation and drug development are hindered, in part, by the lack of objective disease markers.

This is a multi-center trial to validate a potential biomarker for ALS, known as intermuscular coherence (IMC-βγ). IMC measures the correlation in the activity of two muscles during a simple motor task. In a preliminary study we found that patients with ALS have lower IMC than do control subjects. Because measuring IMC is quick, non-invasive, painless, and only requires equipment readily available in standard clinical neurophysiology labs, if validated it would be an important biomarker for ALS.

ELIGIBILITY:
Inclusion Criteria:

* AIM 1: Patients with arm or leg weakness, spastic gait, muscle wasting and/or fasciculations (muscle twitching), dysphagia (difficulty swallowing), dysarthria (difficulty speaking), shortness of breath, hyperreflexia or pathological reflexes, or findings of muscle denervation in previous needle electromyography (EMG) studies.
* AIM 2: Subjects between 20 and 90 years of age.
* AIM 3: Subjects will be selected from among Aim 1 patients who carry an Awaji (without IMC) category of Possible, Probable, or Definite ALS.

Exclusion Criteria:

* AIM 1:

  1. Classified as probable or definite ALS by Awaji criteria prior to initial study evaluation
  2. Have significant sensory loss in the weak or spastic limbs
  3. Have significant musculoskeletal or neuropathic pain
  4. Have an inability or are unwilling to provide informed consent
  5. Are unable to perform the study-related task
  6. Are taking baclofen or benzodiazepines
  7. Have a known non-ALS cause for symptoms
* AIM 2:

  1. Have a history of neurological disorders such as stroke, neuropathy, or myopathy
  2. Have significant pain or sensory loss
  3. Are taking baclofen or sedatives such as benzodiazepines
  4. Lack of cognitive ability or willingness to provide informed consent
* AIM 3:

  1. Were unclassified according to the Awaji category or had a defined ALS mimic
  2. Are taking baclofen, sedatives or benzodiazepines.

NOTE: Participation in a therapeutic clinical trial is NOT an exclusion criterion since this study would not interfere with any potential interventions.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: AIM 1: The study population includes patients with symptomatology suggestive of ALS who are referred to neuromuscular clinics at one of the four participating centers.
  AIM 2: All healthy subjects between 20 and 90 years old.
  AIM 3: Patients with suspected ALS who had an initially detectible IMC-βγ.
Sampling Method: Non-Probability Sample
Enrollment: 650 (Estimated)
Dates: Start 2021-03-31 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in the sensitivity for diagnosing ALS when a measure of intermuscular coherence is added to the Awaji criteria. | 5 years
  Aim 1 asks if incorporation of IMC-βγ into the Awaji criteria improves the criteria's sensitivity for diagnosing ALS.

SECONDARY OUTCOMES:
Time to diagnosis of ALS | 5 years
  Aim 1 asks if incorporation of IMC-βγ into the Awaji criteria reduces the time to diagnosis of ALS.
Rate of ALS disease progression | 5 years
  Aim 3 asks whether changes in the magnitude of IMC-βγ measured over many months varies with ALS disease progression in patients.

CONTACTS AND LOCATIONS:
Overall Officials: Kourosh Rezania, MD, Principal Investigator — University of Chicago
Locations (4):
- United States (4):
  - University of California Center for Clinical Research, Irvine, California
  - University of Miami Miller School of Medicine, Miami, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Washington University Medical Center, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Issa NP, Frank S, Roos RP, Soliven B, Towle VL, Rezania K. Intermuscular coherence in amyotrophic lateral sclerosis: A preliminary assessment. Muscle Nerve. 2017 Jun;55(6):862-868. doi: 10.1002/mus.25426. Epub 2017 Feb 3. PMID 27699797
- See also: Intermuscular coherence in amyotrophic lateral sclerosis: A preliminary assessment — https://pubmed.ncbi.nlm.nih.gov/27699797/